CLINICAL TRIAL: NCT06540040
Title: A Comparative Study to Assess the Efficacy of Postoperative Dressing in the Prevention of Early Surgical Site Complication and Facilitation of Early Mobilization After Orthopaedic Surgeries on Hip and Knee
Brief Title: Comparative Efficacy of Advanced and Traditional Wound Dressings in Post-Operative Orthopedic Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nidhi Srivastava (Other)
Responsible Party: Sponsor-Investigator, Nidhi Srivastava, Ortho Matron, Base Hospital Delhi Cantt
Organization: Base Hospital Delhi Cantt (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 88/2022
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Orthopaedics Wound Dressings
Keywords: wound healing; surgical wound infection; Randomised Controlled Tmrial; Patient comfort; Pain management
MeSH Terms: conditions — Surgical Wound Infection; Agnosia

STUDY DESIGN:
Intervention Model Description: ### Model Description
  **Parallel Assignment**: This study employs a parallel assignment model, where participants are randomly allocated to one of four intervention groups. Each group receives a distinct type of wound dressing post-operatively. The outcomes are measured and compared across these groups to evaluate the efficacy of each dressing type. The interventions include Aquacel Ag, OPSITE, MEPILEX POST OP BORDER, and traditional gauze-based dressings. This model allows for a direct comparison of the different interventions in a controlled manner.
Masking Description: his study is an open-label trial, meaning that there is no masking. All parties involved in the study, including participants, care providers, investigators, and outcome assessors, are aware of the type of dressing each participant receives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Aquacel Ag (Experimental): Participants in this group will receive Aquacel Ag, a Hydrofibre wound dressing consisting of non-woven sodium carboxymethylcellulose fibres integrated with ionic silver. This dressing is designed to provide a moist wound environment and has antimicrobial properties to help reduce the risk of infection. The dressing will be applied post-operatively and changed as per the standardized protocol.
  Interventions: Device: Aquacel Ag
- OPSITE (Experimental): Participants in this group will receive OPSITE, a transparent waterproof cotton pad with a high Moisture Vapour Transmission Rate. This dressing is intended to provide a protective barrier while allowing moisture vapor to escape, helping to maintain an optimal wound healing environment. The dressing will be applied post-operatively and changed according to the standardized protocol.
  Interventions: Device: OPSITE
- MEPILEX POST OP BORDER (Experimental): Participants in this group will receive MEPILEX POST OP BORDER, a 4-layer foam dressing with flex technology. This advanced dressing is designed to provide superior absorption and conformability, helping to manage exudate and protect the wound site. The dressing will be applied post-operatively and changed as per the standardized protocol.
  Interventions: Device: MEPILEX POST OP BORDER
- Traditional Dressing (Active Comparator): Participants in this group will receive traditional wound dressings consisting of gauze pieces, surgical pads, and porous paper adhesive strips. This type of dressing is commonly used in post-operative care to absorb exudate and protect the wound site. The dressing will be applied post-operatively and changed according to the standardized protocol.
  Interventions: Device: Traditional Dressing

INTERVENTIONS:
Device: Aquacel Ag — Aquacel Ag is a Hydrofibre wound dressing composed of non-woven sodium carboxymethylcellulose fibers integrated with ionic silver. It is designed to provide a moist wound environment and has antimicrobial properties to help reduce the risk of infection. The dressing will be applied post-operatively and changed according to a standardized protocol.
  Other Names: Hydrofibre wound dressing with ionic silver
  Arms: Aquacel Ag
Device: OPSITE — OPSITE is a transparent waterproof dressing with a high Moisture Vapour Transmission Rate. It is intended to provide a protective barrier while allowing moisture vapor to escape, maintaining an optimal wound healing environment. The dressing will be applied post-operatively and changed according to a standardized protocol.
  Other Names: Transparent waterproof cotton pad
  Arms: OPSITE
Device: MEPILEX POST OP BORDER — MEPILEX POST OP BORDER is a 4-layer foam dressing designed with flex technology for superior absorption and conformability. It helps manage exudate and protects the wound site. The dressing will be applied post-operatively and changed according to a standardized protocol.
  Other Names: 4-layer foam dressing with flex technology
  Arms: MEPILEX POST OP BORDER
Device: Traditional Dressing — Traditional dressing involves the use of gauze pieces, surgical pads, and porous paper adhesive strips. This type of dressing is commonly used in post-operative care to absorb exudate and protect the wound site. The dressing will be applied post-operatively and changed according to a standardized protocol.
  Other Names: Gauze pieces, surgical pads, and porous paper adhesive strips
  Arms: Traditional Dressing

SUMMARY:
Title: Comparative Efficacy of Advanced and Traditional Wound Dressings in Post-Operative Orthopedic Care: A Randomized Controlled Trial

Objective:

The primary objective of this study is to evaluate and compare the efficacy of advanced wound dressings versus traditional gauze-based dressings in post-operative orthopedic care. The study aims to assess various parameters including patient comfort, pain management, ease of application, exudate management, and the incidence of early surgical site complications.

DETAILED DESCRIPTION:
Title: Comparative Efficacy of Advanced and Traditional Wound Dressings in Post-Operative Orthopedic Care: A Randomized Controlled Trial

Brief Summary:

This study aims to compare the efficacy of advanced wound dressings with traditional gauze-based dressings in post-operative orthopedic care. The study evaluates patient comfort, pain management, ease of application, exudate management, and the incidence of early surgical site complications.

Study Type: Interventional (Clinical Trial)

Study Design: Randomized Controlled Single-Centre Open-Label Study

Primary Purpose: Treatment

Study Start Date: August 10, 2022

Study Completion Date: December 10, 2022

Primary Completion Date: December 10, 2022

Estimated Enrollment: 320 participants

Intervention Model: Parallel Assignment

Masking: None (Open Label)

Interventions:

Participants undergoing orthopedic surgical procedures were randomized into four groups:

Group A: Aquacel Ag (Hydrofibre wound dressing with ionic silver) Group B: OPSITE (Transparent waterproof cotton pad with high Moisture Vapour Transmission Rate) Group C: MEPILEX POST OP BORDER (4-layer foam dressing with flex technology) Group D: Traditional dressing with gauze pieces, surgical pads, and porous paper adhesive strips

Objectives:

To assess the incidence of early surgical site complications such as blisters, infection, maceration, rashes, redness, swelling, and dehiscence at days 3, 7, and 14.

To determine the pain and discomfort experienced by patients during dressing changes using a visual analog scale.

To evaluate the ability to perform activities of daily living comfortably. To assess nurses' ease of application and removal of the dressings.

Outcome Measures:

Primary Outcome Measures: Incidence of surgical site complications at days 3, 7, and 14.

Secondary Outcome Measures: Pain levels during dressing changes, comfort and mobility in daily activities, ease of application and removal of the dressings, and patient satisfaction.

Data Collection Methods:

Data were collected using a semi-structured questionnaire validated by experts. The questionnaire included a wound assessment checklist, a 10-point Likert scale for patient comfort and mobility, a Visual Analog Scale for pain, and a rating scale for nurses' ease of application and removal.

Statistical Analysis:

Categorical variables were presented as numbers and percentages. Continuous variables were presented as mean ± SD and median values. Data normality was checked using the Kolmogorov-Smirnov test. Quantitative variables were analyzed using ANOVA and Kruskal-Wallis test with post hoc tests as appropriate.

Qualitative variables were analyzed using the Chi-Square test or Fisher's exact test for cells with expected values less than 5.

A p-value of less than 0.05 was considered statistically significant.

Ethics and Registration:

Detailed Description:

This study evaluates the comparative efficacy of different wound dressings used in post-operative orthopedic care. The focus is on advanced dressings such as Aquacel Ag, OPSITE, and MEPILEX POST OP BORDER, compared to traditional gauze-based dressings. The study measures various parameters including patient comfort, pain during dressing changes, ease of application and removal by nurses, and management of wound exudate. Data were collected at three time points: days 3, 7, and 14 post-surgery. The results aim to provide insights into the best practices for post-operative wound management in orthopedic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years Undergoing orthopedic surgical procedures, elective or trauma, with a surgical wound size of more than 5 cm Provided informed consent

Exclusion Criteria:

* Open fractures Revision surgeries Established infections Ongoing pharmacological anticoagulation prophylaxis Predisposing skin conditions Known allergy or hypersensitivity to any of the constituents of the dressings Any associated systemic injury precluding early mobilization Unwillingness to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Early Surgical Site Complications | Day 3, Day 7, Day 14 post-surgery
  The primary outcome measure will be the incidence of early surgical site complications, including blisters, skin margin infection, maceration, rashes, redness, swelling, and wound dehiscence. These complications will be assessed at three time points: day 3, day 7, and day 14 post-surgery.

SECONDARY OUTCOMES:
Pain Levels During Dressing Changes | Day 3, Day 7, Day 14 post-surgery
  Pain levels experienced by patients during dressing changes will be assessed using a Visual Analog Scale (VAS) from 0 to 10, where 0 corresponds to no pain and 10 corresponds to unbearable pain. This will be measured at day 3, day 7, and day 14 post-surgery.
Patient Comfort and Mobility | Day 3, Day 7, Day 14 post-surgery
  Patient comfort and ability to perform activities of daily living will be assessed using a 0-to-10-point scale, where 0 indicates absolute discomfort and 10 indicates no limitation due to the dressing. This will be measured at day 3, day 7, and day 14 post-surgery.
Nurses' Ease of Application and Removal of Dressings | Day 3, Day 7, Day 14 post-surgery
  Nurses will rate the ease of application and removal of the dressing using a 0-to-10-point scale, considering factors such as time taken, difficulty, and any issues encountered during the process. This will be measured at day 3, day 7, and day 14 post-surgery.
Patient Satisfaction Levels | Day 14 post-surgery
  Patient satisfaction with the dressing will be assessed using a structured questionnaire. This will be measured at day 14 post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Amresh Ghai, MS (Ortho), Study Director — Base Hospital Delhi Cantt
Locations (1):
- Base Hospital Delhi cantt, New Delhi, India

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers.

REFERENCES:
- [Derived] Srivastava N, Manisha, Ghai A, Goyal M, Kumar M, Kumar M. Comparative efficacy of advanced and traditional wound dressings in post-operative orthopaedic care for hip and knee surgeries: A randomized controlled trial. J Clin Orthop Trauma. 2025 Feb 12;63:102933. doi: 10.1016/j.jcot.2025.102933. eCollection 2025 Apr. PMID 40070522